CLINICAL TRIAL: NCT05882474
Title: Correlation Between Level of Partial Pressure of Carbon Dioxide and Respiratory Effort in Patients With COVID-19 Undergoing Pressure Support Ventilation With Extracorporeal Membrane Oxygenation
Brief Title: Correlation Between PaCO2 and Respiratory Effort in Patients With COVID-19 With Extracorporeal Membrane Oxygenation
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-PUMCH-A-216-2
Record Dates: First submitted 2023-05-27; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation Complication; Respiratory Effort-Related Arousal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- baseline group: PaCO2 35~40mmHg
- High-CO2 group: PACO2 increases by 5-10mmHg compared to baseline value and >40mmHg
  Interventions: Device: PaCO2

INTERVENTIONS:
Device: PaCO2 — Level of partial pressure of carbon dioxide
  Groups: High-CO2 group

SUMMARY:
Excessive respiratory effort may cause self-inflicted lung injury (SILI) and inspiratory muscle injuries , stimulate desynchronization between the patient and ventilator , and worsen the perfusion of extrapulmonary organs . Appropriate respiratory drive and effort should be maintained during the treatment of patients with respiratory failure . In contrast, respiratory drive and effort are commonly increased in patients with COVID-19 pneumonia , and this phenomenon may persist in critically ill patients with COVID-19, even after receiving venovenous ECMO (vv-ECMO) support, owing to low pulmonary compliance and a high systemic inflammatory state .

To reduce respiratory effort and drive, ICU physicians often administer high doses of sedative drugs, analgesics, and muscle relaxants. The prolonged use of high doses of these drugs can cause loss of the spontaneous cough reflex, which in turn impairs sputum drainage and eventually worsens pulmonary consolidation and lung infections.

As the partial pressure of carbon dioxide in arterial blood (PaCO2) could affect the respiratory drive from the respiratory center (1), it has been shown that altering different levels of extracorporeal carbon dioxide removal in patients undergoing ECMO recovering from acute respiratory distress syndrome (ARDS) could alter respiratory drive. We hope to find a more appropriate target for maintaining PaCO2 to control respiratory effort in patients with COVID-19 undergoing ECMO.

DETAILED DESCRIPTION:
A stable environment was maintained during the study to avoid stress and abrupt stimulation.

Before the start of the study, sedative drugs were titrated to Richmond agitation sedation scale values of -3 to -2, an assisted breathing mode trial was conducted, and support pressure level were adjusted to achieve tidal volume < 6 mL/kg. The ECMO GF was adjusted to achieve stable baseline conditions, defined as PaCO2 < 40 mmHg, respiratory rate < 25 bpm, and peak airway pressure < 25 cm H2O. PEEP, fraction of inspired oxygen, pressure support ventilation (PSV), ECMO blood flow, and dose of vasoconstrictors, sedatives, and analgesics remained unchanged throughout the study.

The study protocol was initiated when the baseline parameters s were stable. The baseline parameters, including ventilation settings, arterial and arterial blood gas analysis, hemodynamics, and indicators of respiratory effort were measured in the baseline group. Then, the ECMO GF was modified to 50% of the baseline, and etCO2 values were monitored. ECMO GF was adjusted at 5-min intervals (increasing or decreasing by 0.5 L/min each time) until etCO2 stabilized at a level 5-10 mmHg higher than the baseline. After 20 min, the parameters were measured for the second time in the high-CO2 group (Figure 1).

The study was stopped if the heart rate (HR) was > 140 beats/min and/or respiratory rate was > 40 bpm and/or systolic blood pressure > 180 mmHg and/or patients experienced anxiety or diaphoresis.

ELIGIBILITY:
Inclusion Criteria:

Patients with COVID-19 who had undergone ECMO and pressure support ventilation (PSV) via tracheal intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted in the ICU of Peking Union Medical College Hospital in China. Patients with COVID-19 who had undergone ECMO and pressure support ventilation (PSV) via tracheal intubation between December 2022 and March 2023 were considered eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Pressure muscle index | Not exceeding 1 hour
  During the pressure support mode, the inspiratory hold button was pressed and a physician performed an end-inspiratory occlusion maneuver. After a certain period, the patient completely stopped inspiratory effort. The difference between the end-inspiratory obstructive plateau pressure and pre-obstructive airway pressure (Paw) was used to estimate the patient's inspiratory effort and referred to as Pressure muscle index
airway pressure swing during occlusion | Not exceeding 1 hour
  is defined as the swing in the Paw generated by the force of the respiratory muscle under assisted ventilation when the airway is temporarily blocked (3). The expiratory airway occlusion of the ventilator was performed at random intervals during each recording. Each occlusion persisted for a single breath, as verified by the normal recovery of Paw. The maximum deviation of Paw from positive end-expiratory pressure (PEEP) during each occlusion was documented as airway pressure swing during occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Basic characteristics, vital signs, monitoring indicators, and other information of enrolled patients